CLINICAL TRIAL: NCT04453488
Title: Double-blind, Randomized, Placebo-controlled Clinical Trial to Evaluate the Efficacy of the RUTI® Vaccine to Prevent SARS-CoV-2 Infection
Brief Title: Clinical Trial to Evaluate the Efficacy of RUTI® Against SARS-COV-2 Infection (COVID-19) in Healthcare Workers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RUTICOVID19
Record Dates: First submitted 2020-06-30; First posted 2020-07-01 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Covid-19; Sars-CoV2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RUTI® vaccine (Experimental): Participants will receive two dose of RUTI® vaccine at the baseline visit and after 2 weeks +/- 3 days, which will be administered subcutaneously in the deltoid region at a dose of 25 µg of fragmented, purified and liposomed heat-inactivated Mycobacterium tuberculosis bacilli in an injection volume of 0.3 mL.
  Interventions: Biological: RUTI® vaccine
- Placebo (Placebo Comparator): Participants will receive two dose of physiological serum will be administered subcutaneously in the deltoid region at the baseline visit and after 2 weeks +/- 3 days.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RUTI® vaccine — Each dose of the RUTI® vaccine contains 25 µg of fragmented, purified and liposomed heat-inactivated Mycobacterium tuberculosis bacilli.
  Arms: RUTI® vaccine
Biological: Placebo — Physiological serum, 0.9% NaCl, will be used as a placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of RUTI® vaccine preventing SARS-CoV-2 infection (COVID-19) in healthcare workers.

DETAILED DESCRIPTION:
The aim of this study is to assess the efficacy of RUTI® vaccine preventing SARS-CoV-2 infection (COVID-19) in healthcare workers. The study will include a comparison between placebo and RUTI® vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the Informed Consent before initiating the selection procedures.
2. Healthcare system workers working in contact with subjects potentially infected with SARS-CoV-2.
3. People ≥ 18 years.
4. Willingness to meet the requirements of the protocol.
5. Negative Rapid Serological Test of SARS-CoV-2
6. The participant must agree to use effective contraceptive methods during the study period, in case of childbearing age.

Exclusion Criteria:

1. Previous SARS-CoV-2 infection
2. Pregnancy. Pregnancy test will be performed in case of doubt.
3. Breastfeeding.
4. Suspected of active viral or bacterial infection.
5. Symptoms compatible with COVID-19, despite a negative polymerase chain reaction (PCR) test.
6. Vaccination in the last 4 weeks or planned vaccination during the study period, except for influenza vaccine.
7. Participation in a research that requires experimental intervention (does not include observational studies) in the previous month before signing the Consent or during the study.
8. Severely immunocompromised people. This exclusion category includes:

   1. Subjects with human immunodeficiency virus (HIV-1).
   2. Neutropenic subjects with less than 500 neutrophils / mm3.
   3. Subjects with solid organ transplantation.
   4. Subjects with bone marrow transplantation.
   5. Subjects undergoing chemotherapy.
   6. Subjects with primary immunodeficiency.
   7. Severe lymphopenia with less than 400 lymphocytes / mm3.
   8. Treatment with any anti-cytokine therapy.
   9. Oral treatment with steroids, defined as daily doses of 10 mg prednisone or equivalent for more than 3 months.
9. Malignancy, or active solid or non-solid lymphoma from the previous two years.
10. BCG vaccination in the last 1year.
11. Soy allergy.

12 Chloroquine or hydroxychloroquine administration in the last two weeks.

13. Direct involvement in the design or execution of the RUTICOVID19 clinical trial.

14 Retirement, transfer, long-term leave (> 1 month) due to scheduled surgery or any other event that makes it impossible to work in person at your health center during the months following the recruitment to the study.

15. Employee at the health center <22 hours per week.

16. Do not have a smartphone.

17. Detection by the researcher of lack of knowledge or willingness to participate and comply with all requirements of the protocol.

18. Any other findings that, at the discretion of the researcher, may compromise compliance with the protocol or that may influence significantly the interpretation or the results of the effects of the vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2020-07-30 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Documented cumulative incidence of SARS-CoV-2 infection | Up to 4 months
  % positive serology at the end of the study or positive PCR test in the course of routine clinical practice

SECONDARY OUTCOMES:
Sick leave for SARS-CoV-2 | Up to 4 months
  Number of days of documented sick leave for SARS-CoV-2
Days off work due to the quarantine | Up to 4 months
  The number of days off work due to the quarantine imposed as a consequence to have acute respiratory symptoms, fever or infection documented by SARS-CoV-2
Quarantine imposed by close contact outside the center with SARS-CoV-2 positive | Up to 4 months
  Number of days of quarantine imposed by close contact outside the center with SARS-CoV-2 positive
Professional category | Up to 4 months
  Number of MD, nursing, personnel management and services, etc.
Fever | Up to 4 months
  Number of days of self-reported fever (≥38 ºC)
Incidence of self-reported acute respiratory symptoms | Up to 4 months
  Cumulative incidence of self-reported acute respiratory symptoms
Days of self-reported acute respiratory symptoms | Up to 4 months
  Number of days of self-reported acute respiratory symptoms
Incidence of pneumonia | Up to 4 months
  Number of participants with pneumonia confirmed by X-ray
Incidence of death from SARS-CoV-2 infection | Up to 4 months
  Cumulative incidence of death from documented SARS-CoV-2 infection
Incidence of admissions to Intensive Care Unit (ICU) | Up to 4 months
  Cumulative incidence of admissions to intensive care unit for documented SARS-CoV-2 infection
Days in ICU | Up to 4 months
  Number of days admitted to the ICU for documented SARS-CoV-2 infection
Incidence of mechanical ventilation | Up to 4 months
  Cumulative incidence of need for mechanical ventilation due to documented SARS-CoV-2 infection
Incidence of hospital admissions | Up to 4 months
  Cumulative incidence of hospital admissions for documented SARS-CoV-2 infection
Days of hospitalization | Up to 4 months
  Number of days of hospitalization for documented SARS-CoV-2 infection
Incidence of SARS-CoV-2 antibodies | Final visit
  Incidence of SARS-CoV-2 antibodies at the end of the study period
Types of antibodies detected | Final visit
  Frequency and levels of immunoglobulin IgG and immunoglobulin IgM
Levels of SARS-CoV-2 antibodies | Final visit
  Levels of SARS-CoV-2 antibodies at the end of the study period

OTHER OUTCOMES:
AEs | Up to 4 months
  All adverse events reported by the subjects, both serious and non-serious, will be collected. All events related to a SARS-CoV-2 infection will be exempted from collection as part of the associated symptoms.
SAEs | Up to 4 months
  All those Adverse Events that lead to hospitalization of the patient, that endanger his life or cause or may cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Pere-Joan Cardona, MD, PhD, Study Chair — IGTP
Locations (2):
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol UBP Riscos Laborals, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: No